CLINICAL TRIAL: NCT02583464
Title: Bioequivalence Study of Two Formulations With the Association of Tenofovir 300 mg and Emtricitabine 200 mg.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BE-TNF-EMT
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test-Reference (Experimental): A new formulation containing a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg (T) followed by a branded formulation (R).
  Interventions: Drug: Tenofovir disoproxil fumarate and emtricitabine
- Reference-Test (Experimental): A branded formulation containing a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg (R) followed by a new formulation (T).
  Interventions: Drug: Tenofovir disoproxil fumarate and emtricitabine

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate and emtricitabine — Two period administration of a formulation containing a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg.

SUMMARY:
Objective: To evaluate the relative bioavailability of a new formulation containing a combination of emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg (T) and compare this formulation with the branded formulation (R) to meet regulatory criteria for marketing the test product in Argentina.

DETAILED DESCRIPTION:
A randomized-sequence, open-label, two-period crossover study was conducted on 24 healthy Caucasian volunteers in a fasting state. A single oral dose of either T or R formulations was followed by a 7-day washout period. Blood samples were collected at baseline and 0.25, 0.50, 0.75, 1, 1.25, 1.5 2, 2.5, 3, 4, 7, 12, 24 and 48 h after administration. Emtricitabine and tenofovir concentrations were determined using a validated LC (liquid chromatography) - MS (mass spectrometry) / MS method. Adverse events were monitored based on clinical parameters and volunteer reports.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both sexes between 21 and 55 years.
2. Subjects with body mass index (BMI) between 19 and 27 kg / m².
3. Subjects whose complementary tests (ECG, blood and urine) are within normal and / or clinically insignificant according to the judgment of the investigator. Women of childbearing age should have a negative pregnancy test and use a reliable method of contraception during the study (IUD or condoms)
4. Subjects with systolic blood pressure between 110 mmHg and 139 mmHg; diastolic pressure between 70 mmHg and 89 mmHg; heart rate between 50 and 90 beats per minute.
5. Subjects who signed informed consent.

Exclusion Criteria:

1. Background of clinically significant allergies (except untreated asymptomatic seasonal allergies), drug hypersensitivity and / or hypersensitivity to any component of the formulations studied.
2. Drop of more than 20 mmHg in systolic blood pressure or more than 10 mmHg diastolic pressure in the first 3 minutes of postural change.
3. Active smoker more than 10 cigarettes / day.
4. Pregnant or lactating women.
5. Current clinical evidence of severe digestive disorders, surgery of the digestive tract (except appendectomy).
6. Current clinical evidence of kidney disease.
7. Current evidence of liver disorders
8. Current clinical evidence of respiratory and heart diseases.
9. The presence of diabetes mellitus, thyroid dysfunction or other endocrine disorder.
10. Evidence of gastroduodenal disease.
11. Current presence of any malignancy.
12. History of abuse or addiction to drugs or alcohol during the past three years.
13. Participation in a clinical trial within the last three months.
14. Use of any drug within fourteen days before the start of the study.
15. Subject donated or suffered blood loss during the last twelve weeks before the start of the study, or intends to donate blood within three months of the completion of the study.
16. Excessive drinking of tea, cocoa, mate, coffee and / or beverages containing caffeine (> 5 cups / day) or wine (> 0.5 L / day) or alcohol (> 50 ml / day).
17. ECG abnormalities.
18. Positive serology for HIV, hepatitis B or hepatitis C.
19. Women who are not using effective contraception (IUD, condom)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 48 hours
Area Under the Curve [AUC] | 48 hours

SECONDARY OUTCOMES:
Adverse events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Di Girolamo, MD, Principal Investigator — Centro de la Asociación Mutual de Profesionales del Hospital Italiano
Locations (1):
- Laboratorio Elea SACIFyA, Capital Federal, Buenos Aires, Argentina